CLINICAL TRIAL: NCT05979415
Title: A Randomized, Double-Blind, to Evaluate the Efficacy and Safety of Staccato Apomorphine (AZ-009) in Patients With Parkinson's Disease Experiencing OFF Episodes
Brief Title: Study to Evaluate the Efficacy and Safety of Staccato Apomorphine (AZ-009) in Patients With Parkinson's Disease Experiencing OFF Episodes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative decision
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Collaborators: Peachtree BioResearch Solutions Inc. (Unknown); DSG, Inc (Unknown); ISS, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMDC 009-201
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
Keywords: OFF episode
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Staccato Apomorphine (Active Comparator): 1mg, 2mg, 3mg, 4mg
  Interventions: Drug: Apomorphine Cartridge
- Staccato Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Apomorphine Cartridge

INTERVENTIONS:
Drug: Apomorphine Cartridge — Staccato Cartridge
  Other Names: placebo

SUMMARY:
This study will be conducted with In-clinic visits and treatment at home for each patient with established Parkinson's disease (PD) experiencing daily OFF episodes.

DETAILED DESCRIPTION:
The purpose of this protocol is to establish the safety, tolerability, and efficacy of AZ-009 compared to placebo in patients with established PD experiencing daily OFF episodes.

Patients between the ages of 30 and 85 with a clinical diagnosis of established PD who experience motor fluctuation and have recognizable OFF periods are eligible for participation in this study. The patients will be classified as Modified Hoehn & Yahr stage II-IV in the ON state and have clear, self-described daily motor fluctuations while on oral l-dopa or Carbidopa (with or without adjunctive PD therapy).

This study will be conducted in approximately 50 patients, with up to 8 Open-Label titration in-clinic visits with treatment at home between visits. This is followed by Double Blind which includes a 13 day treatment at home period, and an in-clinic visit and an End of Study/Early Termination visit for each patient with established Parkinson's disease (PD) experiencing daily OFF episodes.

ELIGIBILITY:
Inclusion Criteria:

* 1. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted.

  2. Willing and able to travel to the clinical research center and adhere to the overall study visit schedule, procedures, and other protocol requirements.

  3. Male or female between the ages of 30 and 85 (inclusive). 4. Body weight ≥ 50 kg. 5. Willing to abstain from alcohol for 6 hours prior to a study visit and minimize alcohol use throughout the study duration.

  6. Have a clinical diagnosis of PD; with fulfillment of Steps 1 and 2 of the UK Parkinson's Disease Brain Bank Criteria.

  7. Optimized and stabilized on oral dopaminergic therapy including levodopa at least 3 times daily and in combination with decarboxylase inhibitor at least 30 days prior to screening.

  8. Classified as Modified Hoehn & Yahr stage II-IV in the ON state at Visit 1. 9. Have an MDS-UPDRS III score of at least 30 in the OFF state prior to the L-dopa challenge at Visit 2.

  10. Experience self-described motor fluctuations (confirmed by the Motor Fluctuation Questionnaire at Screening) with recognizable OFF periods while on optimized oral l-dopa or dopamine agonist therapy.

  11. Experience at least 2 hours of OFF time per day and show responsiveness to levodopa (defined by a ≥ 30% reduction in MDS-UPDRS III score compared to pre-dose) at Visit 2.

  12. Female subjects, who are not pregnant or breastfeeding, and one of the following conditions applies: 13. Surgically sterile (including bilateral tubal ligation) for at least 3 months prior to screening.
  * Postmenopausal, defined as 1 of the following:
  * Last menstrual sequence greater than 12 months prior to screening
  * Last menstrual sequence greater than 6 months prior to screening and a serum follicle-stimulating hormone (FSH) concentration > 40 mIU/mL
  * Of childbearing potential (i.e., do not meet the criteria outlined above), patient must:
  * Have a negative urine pregnancy test at Screening and Day -1, as verified by the study doctor prior to starting study therapy.
  * Either commit to true abstinence from heterosexual contact or agree to use, and be able to comply with, effective contraception without interruption with one of the following methods during the study participation up until 30 days after administration of study drug:
  * Oral contraceptive medications; Intra uterine devices; Hormonal implants; Injectable contraceptive medications; Double-barrier methods 14. Male subjects must practice true abstinence from heterosexual contact or, during sexual contact with a pregnant female or a female of childbearing potential, agree to use a condom or have had vasectomy with negative semen analysis and refrain from sperm donation during the duration of the study and up to 90 days after last dose of study drug.

Exclusion Criteria:

* Subjects eligible for enrollment in the study must meet all of the following inclusion criteria and none of the exclusion criteria.

Inclusion Criteria:

1. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted.
2. Willing and able to travel to the clinical research center and adhere to the overall study visit schedule, procedures, and other protocol requirements.
3. Male or female between the ages of 30 and 85 (inclusive).
4. Body weight ≥ 50 kg.
5. Willing to abstain from alcohol for 6 hours prior to a study visit and minimize alcohol use throughout the study duration.
6. Have a clinical diagnosis of PD; with fulfillment of Steps 1 and 2 of the UK Parkinson's Disease Brain Bank Criteria.
7. Optimized and stabilized on oral dopaminergic therapy including levodopa at least 3 times daily and in combination with decarboxylase inhibitor at least 30 days prior to screening.
8. Classified as Modified Hoehn & Yahr stage II-IV in the ON state at Visit 1.
9. Have an MDS-UPDRS III score of at least 30 in the OFF state prior to the L-dopa challenge at Visit 2.
10. Experience self-described motor fluctuations (confirmed by the Motor Fluctuation Questionnaire at Screening) with recognizable OFF periods while on optimized oral l-dopa or dopamine agonist therapy.
11. Experience at least 2 hours of OFF time per day and show responsiveness to levodopa (defined by a ≥ 30% reduction in MDS-UPDRS III score compared to pre-dose) at Visit 2.
12. Female subjects, who are not pregnant or breastfeeding, and one of the following conditions applies:
13. Surgically sterile (including bilateral tubal ligation) for at least 3 months prior to screening.

    * Postmenopausal, defined as 1 of the following:
    * Last menstrual sequence greater than 12 months prior to screening
    * Last menstrual sequence greater than 6 months prior to screening and a serum follicle-stimulating hormone (FSH) concentration > 40 mIU/mL
    * Of childbearing potential (i.e., do not meet the criteria outlined above), patient must:
    * Have a negative urine pregnancy test at Screening and Day -1, as verified by the study doctor prior to starting study therapy.
    * Either commit to true abstinence from heterosexual contact or agree to use, and be able to comply with, effective contraception without interruption with one of the following methods during the study participation up until 30 days after administration of study drug:
    * Oral contraceptive medications; Intra uterine devices; Hormonal implants; Injectable contraceptive medications; Double-barrier methods
14. Male subjects must practice true abstinence from heterosexual contact or, during sexual contact with a pregnant female or a female of childbearing potential, agree to use a condom or have had vasectomy with negative semen analysis and refrain from sperm donation during the duration of the study and up to 90 days after last dose of study drug.

Exclusion Criteria:

1. Previous significant complications from oral dopamine agonist therapy including hospitalization, hallucinations, or any other clinically relevant neuropsychiatric adverse event. Known intolerance to apomorphine.
2. Inhaled or sublingual apomorphine or inhaled l-dopa treatments during the trial.
3. Expected use of Apokyn or Kynmobi during the titration and treatment phase of the study.
4. Participation in earlier AZ-009 clinical trials.
5. Patients with suicidal behavior occurring within the past year or who pose a current suicide risk as determined by the PI or as confirmed at the first Screening Visit, the L-dopa challenge Visit (Visit -2) or Day 1 (Visit 3) by affirmative answer on items 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS).
6. Symptomatic clinically relevant and medically uncontrolled orthostatic hypotension or systolic blood pressure less than 100 mmHg at Screening or Baseline. Orthostatic hypotension is defined as a decrease in systolic blood pressure of 20 mm Hg > or a decrease in diastolic blood pressure > 10 mm Hg, or increase in heart rate > 20 BPM, when standing compared with blood pressure from the supine position.
7. Any clinically significant or unstable medical or psychiatric condition, as determined by the PI, based on a medical evaluation including history, physical examination, vital signs, electrocardiograms (ECGs), and laboratory tests assessed at the screening visit and prior to the first dose of study drug that could compromise the participant's safety or interfere with the completion of this protocol. A patient with a non-clinically significant abnormality or laboratory parameters outside the reference range may continue with the approval of the Investigator.
8. Subjects with a prolonged QT interval corrected for heart rate according to Fridericia's formula (QTcF) of >450 ms for male and >470 ms for female at screening or directly prior to first dosing, or a history of long QT syndrome. Also subjects with a PR interval > 220 msec or QRS duration > 120 msec at screening.
9. Currently taking, or may need treatment with, nitroglycerine
10. Any documented active or suspected or history of malignancy within 5 years prior to Visit 1, except appropriately treated basal cell carcinoma.
11. Active hallucinations or history of hallucinations in the past 3 months. Any significant medical condition, psychiatric illness, current major uncontrolled depression or bipolar disease, or history of depression that could, in the investigator's opinion, compromise the subject's safety or interfere with the completion of this protocol.
12. Dementia indicated by MMSE <24 at Screening.
13. History of clinically significant central nervous system (e.g., seizures), cardiac, pulmonary (e.g., asthma, COPD), metabolic, renal, hepatic, or gastrointestinal (GI) conditions including gastric bypass or other weight loss surgical procedure; or history of such conditions that, in the opinion of the investigator, may place the subject at an unacceptable risk as a participant in this trial, may interfere with the interpretation of safety and/or tolerability data obtained in the trial, or may interfere with the absorption, distribution, metabolism, or excretion of the study drugs.
14. Screening FEV1 < 50% of predicted or FEV1/FVC ratio < 60% in the ON state at Visit 1.
15. Any condition including the presence of laboratory abnormalities, which according to the investigator places the subject at unacceptable risk if he/she were to participate in the study.
16. Aspartate transaminase (AST), alanine transaminase (ALT), gamma-glutamyl transferase (GGT), serum creatinine, or total bilirubin > 1.5 x upper limit of normal (ULN) at screening or prior to the first dose of study drug. An exception may be made for suspected Gilbert's syndrome. These laboratory tests may be repeated once, if they are abnormal on first screening, and if there is a medical reason to believe the results may be inaccurate. If the repeat test is within the reference range, the subject may be included only if the investigator considers that the previous finding will not compromise the subject's safety and will not interfere with the interpretation of safety data.
17. Positive blood screen for human immunodeficiency virus (HIV antibody), hepatitis B virus surface antigen, or hepatitis C virus antibody at screening.
18. History of drug or alcohol abuse within 6 months of screening.
19. Positive drug screen at baseline. May not be exclusionary with a prescription.
20. History of any smoking/vaping (tobacco, cannabinoids) or any tobacco product use within 3 months prior to the study.
21. Participation in a clinical trial and receipt of an investigational medication or a new chemical entity within 30 days, 5 half-lives, if known, or twice the duration of the biological effect of any medication (whichever is longer) prior to the first dose of current study drug.
22. Use of medication that is inhibitor or inducer of CYP450-3A4/5 within 3 days of dosing.
23. Donation of blood, plasma or other blood products or blood collection in excess of 470 mL within 8 weeks prior to dosing.
24. Known sensitivity to any of the study drugs or components thereof, or a history of medication allergy or other allergy that, in the opinion of the investigator, contraindicates study participation.
25. Major surgery within 4 weeks of screening that could interfere with, or for which the treatment might interfere with, the conduct of the study, or that would pose an unacceptable risk to the subject in the opinion of the investigator.
26. Use of 5HT3 antagonists, including antiemetics (e.g., ondansetron, granisetron, dolasetron, palonosetron) and alosetron during the trial.
27. Medications to treat gastroparesis (Antiemetics) or any dopamine antagonist.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
MDS-Unified Parkinson's Disease Rating Scale | at 10, 20, 30 and 45 minutes
  The MDS-UPDRS is a revision of the Unified Parkinson's Disease Rating Scale (UPDRS) and was developed to evaluate various aspects of Parkinson's disease including non-motor and motor experiences of daily living and motor complications.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Movement Disorders Center of Arizona, Scottsdale, Arizona
  - Tuscon Neuroscience Research (M3 Wake Research), Tucson, Arizona
  - The Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - Cenexel Rocky Mountain Clinical Research, Englewood, Colorado
  - Bradenton Research Center, Inc., Bradenton, Florida
  - Holy Cross Health, Fort Lauderdale, Florida
  - Visionary Investigators Network, Miami, Florida
  - Parkinson's Disease Treatment Center of Southwest Florida, Port Charlotte, Florida
  - CenExel iResearch Atlanta (Decatur), Decatur, Georgia
  - Quest Research Institute, Farmington Hills, Michigan
  - Accellacare of Piedmont Healthcare, Statesville, North Carolina
  - KCA Neurology, (Part of Ki Health Partners, LLC), Franklin, Tennessee
  - Lone Star Neurology, (Part of Ki Health Partners, LLC), Frisco, Texas

IPD SHARING:
Plan to Share IPD: No